CLINICAL TRIAL: NCT06468436
Title: Effect of Dexmedetomidine-Esketamine Combination for Sedation and Analgesia on Delirium in ICU Patients With Mechanical Ventilation: A Multicenter Randomized Trial
Brief Title: Dexmedetomidine-Esketamine Combination for Sedation and Analgesia in ICU Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Collaborators: Peking University International Hospital (Other); Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor and Chairman, Department of Anesthesiology, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2024-239
Record Dates: First submitted 2024-06-15; First posted 2024-06-21 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Aged; Intensive Care Units; Ventilators, Mechanical; Dexmedetomidine; Esketamine; Delirium
Keywords: Aged; Intensive Care Units; Ventilators, Mechanical; Dexmedetomidine; Esketamine; Delirium
MeSH Terms: conditions — Delirium | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexmedetomidine-Esketamine Combination (Experimental): Sedation-analgesia is provided with dexmedetomidine-esketamine combination for up to 14 days or until discharge from the ICU. The formulation consists of dexmedetomidine 200 μg/2 ml and esketamine 100 mg/4 ml, diluted with normal saline to a total volume of 50 ml, resulting in a dexmedetomidine concentration of 4 μg/ml and an esketamine concentration of 2 mg/ml.
  Interventions: Drug: Dexmedetomidine-Esketamine Combination
- Dexmedetomidine (Active Comparator): Sedation-analgesia is provided with dexmedetomidine for up to 14 days or until discharge from the ICU. The formulation consists of dexmedetomidine 200 μg/2 ml, diluted with normal saline to a total volume of 50 ml, resulting in a dexmedetomidine concentration of 4 μg/ml.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine-Esketamine Combination — For patients with invasive ventilation, nighttime sedation (20:00-06:00) is provided with an initial infusion rate of [0.05×kg] ml/h which is increased by [0.025×kg] ml/h every 10 min, until the Richmond Agitation-Sedation Scale (RASS) reaches -2 to -1, maximal infusion rate reaches [0.175×kg] ml/h, or adverse reactions occur. Daytime sedation (06:00-20:00) is provided as above when considered necessary by the ICU physicians, with a target RASS score of -2 to +1.
  For patients with non-invasive ventilation (including high-flow nasal oxygenation) or without assisted ventilation, nighttime sedation (20:00-06:00) is provided with an initial infusion rate of [0.0125×kg] ml/h which is increased by [0.0125×kg] ml/h every 10 min, until the RASS reaches -1, maximal infusion rate reaches [0.05×kg] ml/h, or adverse reactions occur. Daytime sedation (06:00-20:00) is typically not required but is provided when considered necessary by the ICU physicians, with a target RASS score of -1 to +1.
  Other Names: Dexmedetomidine hydrochloride; Esketamine hydrochloride
  Arms: Dexmedetomidine-Esketamine Combination
Drug: Dexmedetomidine — For patients with invasive ventilation, nighttime sedation (20:00-06:00) is provided with an initial infusion rate of [0.05×kg] ml/h which is increased by [0.025×kg] ml/h every 10 min, until the Richmond Agitation-Sedation Scale (RASS) reaches -2 to -1, maximal infusion rate reaches [0.175×kg] ml/h, or adverse reactions occur. Daytime sedation (06:00-20:00) is provided as above when considered necessary by the ICU physicians, with a target RASS score of -2 to +1.
  For patients with non-invasive ventilation (including high-flow nasal oxygenation) or without assisted ventilation, nighttime sedation (20:00-06:00) is provided with an initial infusion rate of [0.0125×kg] ml/h which is increased by [0.0125×kg] ml/h every 10 min, until the RASS reaches -1, maximal infusion rate reaches [0.05×kg] ml/h, or adverse reactions occur. Daytime sedation (06:00-20:00) is typically not required but is provided when considered necessary by the ICU physicians, with a target RASS score of -1 to +1.
  Other Names: Dexmedetomidine hydrochloride
  Arms: Dexmedetomidine

SUMMARY:
Patients with mechanical ventilation in the intensive care unit (ICU) often develop anxiety and agitation, sleep distuebances, and delirium. Delirium occurrence is associated with worse early and long-term outcomes. Dexmedetomidine and ketamine are recommended for sedation and analgesia in ICU patients, but each may induce side effects. The sedative effects of dexmedetomidine can help mitigate the psychiatric side effects of esketamine. Recent studies showed that dexmedetomidine-esketamine combination improved analgesia and sleep quality without increasing psychiatric side effects. This trial is designed to test the hypothesis that dexmedetomidine-esketamine combination for sedation and analgesia in ICU patients with mechanical ventilation may reduce delirium and improve respiratory recovery.

DETAILED DESCRIPTION:
Patients with respiratory failure or other severe conditions often require non-invasive or invasive mechanical ventilation in the Intensive Care Unit (ICU). The uncomfortable stimulation produced by mechanical ventilation may lead to anxiety and agitation of patients and adverse consequences such as ventilator asynchrony, increased oxygen consumption, stress responses, self-extubation, and potentially prolonged mechanical ventilation. The above factors, together with the ICU environment, underlying illnesses, treatment measures, and painful procedures, often result in sleep disturbances in ICU patients.

Mechanical ventilation, painful stimulation, and sleep disturbances are important risk factors of delirium in ICU patients. Delirium is an acutely occurred brain dysfunction symdrome characteristized with fluctuating disturbances in attention, cognition, and consciousness, and is reported to occur in up to 80% of ICU patients with mechanical ventilation. Delirium occurrence is associated with worse outcomes, including prolonged mechanical ventilation duration, extended ICU and hospital stays, increased healthcare burden and costs, and elevated mortality risk, as well as long-term sequelae including cognitive decline, reduced quality of life, and decreased survival.

Dexmedetomidine is a highly selective α2-adrenergic receptor agonist with sedative, analgesic, and anxiolytic effects. It exerts effects by activating the endogenous sleep-promoting pathways, inducing a state like non-rapid eye movement sleep. Ketamine is a non-competitive N-methyl-D-aspartate (NMDA) receptor antagonist. Esketamine, the more potent enantiomer of ketamine, has a higher affinity for the NMDA receptor and is approximately twice as potent as ketamine, with a lower incidence of adverse effects. Both dexmedetomidine and ketamine are recommended for sedation and analgesia in ICU patients. However, sedative dose dexmedetomidine is associated with bradycardia and hypotension. Even low-dose esketamine can induce psychotropic side effects such as dissociation, hallucinations, and nightmares.

The sedative effects of dexmedetomidine can help mitigate the psychiatric side effects of esketamine. Recent studies showed that dexmedetomidine-esketamine combination improved analgesia and sleep quality without increasing psychiatric side effects. It is hypothesized that dexmedetomidine-esketamine combination for sedation and analgesia in ICU patients with mechanical ventilation may reduce delirium and improve respiratory recovery.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years;
2. Receiving invasive or non-invasive mechanical ventilation in the ICU, with an expected duration ≥24 hours;
3. Require sedation as judged by ICU physicians.

Exclusion Criteria:

1. Pregnant or lactating women;
2. History of schizophrenia, epilepsy, Parkinson's disease, or myasthenia gravis;
3. Unable to communicate due to coma, severe dementia, or language barrier prior to invasive/non-invasive mechanical ventilation;
4. After stroke, hypoxic encephalopathy, traumatic brain injury, or neurosurgery;
5. Comorbid with hyperthyroidism or pheochromocytoma;
6. Left ventricular ejection fraction <30%, sick sinus syndrome, severe sinus bradycardia (heart rate <50 bpm), second-degree or higher atrioventricular block without a pacemaker, or systolic blood pressure <90 mmHg despite use of vasopressors;
7. Severe liver dysfunction (Child-Pugh Class C), severe renal dysfunction (requiring dialysis), or expected survival ≤24 hours;
8. Allergy to dexmedetomidine and/or esketamine, or any other conditions that are considered unsuitable for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1508 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2029-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of delirium within 7 days | Up to 7 days after enrollment
  Delirium is assessed twice daily with the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) or the 3-Minute Diagnostic Assessment for Delirium using the Confusion Assessment Method (3D-CAM) during the 7-day period after enrollment or until hospital discharge. Positive result of delirium assessments at any timepoint is defined as occurrence of delirium.

SECONDARY OUTCOMES:
Days alive without delirium or come during the 7-day period | Up to 7 days after enrollment
  Delirium is assessed twice daily with the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) or the 3-Minute Diagnostic Assessment for Delirium using the Confusion Assessment Method (3D-CAM). Coma is defined as Richmond Agitation Sedation Scale (score ranges from -5 [unarousable] to +4 [combative] and 0 indicates alert and calms) of -4 or -5. Positive results at any timepoint is defined as occurrence of delirium or coma.
Ventilator-free days within 30 days | Up to 30 days after enrollment
  Mechanical ventilation includes both invasive and non-invasive ventilation, but do not include high-flow nasal oxygenation.
Length of stay in the ICU | Up to 30 days after enrollment
  Length of stay in the ICU.
30-day all-cause mortality | Up to 30 days after enrollment
  30-day all-cause mortality.

OTHER OUTCOMES:
Proportion of patients without delirium | Up to 7 days after enrollment
  Delirium is assessed twice daily with the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) or the 3-Minute Diagnostic Assessment for Delirium using the Confusion Assessment Method (3D-CAM) during the 7-day period after enrollment or until hospital discharge.
Proportion of patients without delirium or coma | Up to 7 days after enrollment
  Delirium is assessed twice daily with the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) or the 3-Minute Diagnostic Assessment for Delirium using the Confusion Assessment Method (3D-CAM). Coma is defined as Richmond Agitation Sedation Scale (score ranges from -5 [unarousable] to +4 [combative] and 0 indicates alert and calms) of -4 or -5.
Length of stay in hospital after enrollment | Up to 30 days after enrollment
  Length of stay in hospital after enrollment.
Incidence of major complications within 30 days | Up to 30 days after enrollment
  Major complications are defined as new-onset medical conditions other than delirium that are deemed harmful and require therapeutic intervention, that is grade II or higher on the Clavien-Dindo classification.
Incidence of cognitive dysfunction at 30 days | At 30 days after enrollment
  Cognitive function is assessed with the Montreal Cognitive Assessment-telephone version (T-MoCA; score ranges from 0 to 22, with higher score indicating better cognitive function). A decline of 1 standard deviation (SD) or more from baseline is defined as having cognitive dysfunction.
Quality of life at 30 days | At 30 days after enrollment
  Quality of life is assessed with the World Health Organization Quality of Life brief version (WHOQOL-BREF), a 24-item questionnaire that assesses the quality of life in physical, psychological, and social relationship, and environmental domains. The score ranges from 0 to 100 for each domain, with higher score indicating better function.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (3):
- China (3):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University International Hospital, Beijing, Beijing Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fritsch S, Bickenbach J. [Respiratory Insufficiency: State of the Art - Diagnosis and Therapy]. Anasthesiol Intensivmed Notfallmed Schmerzther. 2018 Feb;53(2):90-101. doi: 10.1055/s-0043-107167. Epub 2018 Feb 9. German. PMID 29426048
- [Background] Hempel G, Simon P, Salz P, Wrigge H. [Respiratory Failure: Innovations in Diagnostics and Therapy]. Anasthesiol Intensivmed Notfallmed Schmerzther. 2018 Feb;53(2):126-140. doi: 10.1055/s-0043-108216. Epub 2018 Feb 9. German. PMID 29426051
- [Background] May AD, Parker AM, Caldwell ES, Hough CL, Jutte JE, Gonzalez MS, Needham DM, Hosey MM. Provider-Documented Anxiety in the ICU: Prevalence, Risk Factors, and Associated Patient Outcomes. J Intensive Care Med. 2021 Dec;36(12):1424-1430. doi: 10.1177/0885066620956564. Epub 2020 Oct 9. PMID 33034254
- [Background] Tate JA, Devito Dabbs A, Hoffman LA, Milbrandt E, Happ MB. Anxiety and agitation in mechanically ventilated patients. Qual Health Res. 2012 Feb;22(2):157-73. doi: 10.1177/1049732311421616. Epub 2011 Sep 9. PMID 21908706
- [Background] Cooper AB, Thornley KS, Young GB, Slutsky AS, Stewart TE, Hanly PJ. Sleep in critically ill patients requiring mechanical ventilation. Chest. 2000 Mar;117(3):809-18. doi: 10.1378/chest.117.3.809. PMID 10713011
- [Background] Hardin KA, Seyal M, Stewart T, Bonekat HW. Sleep in critically ill chemically paralyzed patients requiring mechanical ventilation. Chest. 2006 Jun;129(6):1468-77. doi: 10.1378/chest.129.6.1468. PMID 16778263
- [Background] Honarmand K, Rafay H, Le J, Mohan S, Rochwerg B, Devlin JW, Skrobik Y, Weinhouse GL, Drouot X, Watson PL, McKinley S, Bosma KJ. A Systematic Review of Risk Factors for Sleep Disruption in Critically Ill Adults. Crit Care Med. 2020 Jul;48(7):1066-1074. doi: 10.1097/CCM.0000000000004405. PMID 32433122
- [Background] Gehlbach BK, Chapotot F, Leproult R, Whitmore H, Poston J, Pohlman M, Miller A, Pohlman AS, Nedeltcheva A, Jacobsen JH, Hall JB, Van Cauter E. Temporal disorganization of circadian rhythmicity and sleep-wake regulation in mechanically ventilated patients receiving continuous intravenous sedation. Sleep. 2012 Aug 1;35(8):1105-14. doi: 10.5665/sleep.1998. PMID 22851806
- [Background] Elliott R, McKinley S, Cistulli P, Fien M. Characterisation of sleep in intensive care using 24-hour polysomnography: an observational study. Crit Care. 2013 Mar 18;17(2):R46. doi: 10.1186/cc12565. PMID 23506782
- [Background] Rault C, Sangare A, Diaz V, Ragot S, Frat JP, Raux M, Similowski T, Robert R, Thille AW, Drouot X. Impact of Sleep Deprivation on Respiratory Motor Output and Endurance. A Physiological Study. Am J Respir Crit Care Med. 2020 Apr 15;201(8):976-983. doi: 10.1164/rccm.201904-0819OC. PMID 31810378
- [Background] Finan PH, Goodin BR, Smith MT. The association of sleep and pain: an update and a path forward. J Pain. 2013 Dec;14(12):1539-52. doi: 10.1016/j.jpain.2013.08.007. PMID 24290442
- [Background] Fernandes NM, Nield LE, Popel N, Cantor WJ, Plante S, Goldman L, Prabhakar M, Manlhiot C, McCrindle BW, Miner SE. Symptoms of disturbed sleep predict major adverse cardiac events after percutaneous coronary intervention. Can J Cardiol. 2014 Jan;30(1):118-24. doi: 10.1016/j.cjca.2013.07.009. Epub 2013 Oct 16. PMID 24140074
- [Background] Tobaldini E, Fiorelli EM, Solbiati M, Costantino G, Nobili L, Montano N. Short sleep duration and cardiometabolic risk: from pathophysiology to clinical evidence. Nat Rev Cardiol. 2019 Apr;16(4):213-224. doi: 10.1038/s41569-018-0109-6. PMID 30410106
- [Background] Miner SE, Pahal D, Nichols L, Darwood A, Nield LE, Wulffhart Z. Sleep Disruption is Associated with Increased Ventricular Ectopy and Cardiac Arrest in Hospitalized Adults. Sleep. 2016 Apr 1;39(4):927-35. doi: 10.5665/sleep.5656. PMID 26715226
- [Background] Van Rompaey B, Elseviers MM, Schuurmans MJ, Shortridge-Baggett LM, Truijen S, Bossaert L. Risk factors for delirium in intensive care patients: a prospective cohort study. Crit Care. 2009;13(3):R77. doi: 10.1186/cc7892. Epub 2009 May 20. PMID 19457226
- [Background] Slatore CG, Goy ER, O'hearn DJ, Boudreau EA, O'Malley JP, Peters D, Ganzini L. Sleep quality and its association with delirium among veterans enrolled in hospice. Am J Geriatr Psychiatry. 2012 Apr;20(4):317-26. doi: 10.1097/JGP.0b013e3182487680. PMID 22367162
- [Background] Fadayomi AB, Ibala R, Bilotta F, Westover MB, Akeju O. A Systematic Review and Meta-Analysis Examining the Impact of Sleep Disturbance on Postoperative Delirium. Crit Care Med. 2018 Dec;46(12):e1204-e1212. doi: 10.1097/CCM.0000000000003400. PMID 30222634
- [Background] Fong HK, Sands LP, Leung JM. The role of postoperative analgesia in delirium and cognitive decline in elderly patients: a systematic review. Anesth Analg. 2006 Apr;102(4):1255-66. doi: 10.1213/01.ane.0000198602.29716.53. PMID 16551934
- [Background] Wilson JE, Mart MF, Cunningham C, Shehabi Y, Girard TD, MacLullich AMJ, Slooter AJC, Ely EW. Delirium. Nat Rev Dis Primers. 2020 Nov 12;6(1):90. doi: 10.1038/s41572-020-00223-4. PMID 33184265
- [Background] Igwe EO, Nealon J, O'Shaughnessy P, Bowden A, Chang HR, Ho MH, Montayre J, Montgomery A, Rolls K, Chou KR, Chen KH, Traynor V, Smerdely P. Incidence of postoperative delirium in older adults undergoing surgical procedures: A systematic literature review and meta-analysis. Worldviews Evid Based Nurs. 2023 Jun;20(3):220-237. doi: 10.1111/wvn.12649. Epub 2023 May 2. PMID 37128953
- [Background] Krewulak KD, Stelfox HT, Leigh JP, Ely EW, Fiest KM. Incidence and Prevalence of Delirium Subtypes in an Adult ICU: A Systematic Review and Meta-Analysis. Crit Care Med. 2018 Dec;46(12):2029-2035. doi: 10.1097/CCM.0000000000003402. PMID 30234569
- [Background] Ely EW, Inouye SK, Bernard GR, Gordon S, Francis J, May L, Truman B, Speroff T, Gautam S, Margolin R, Hart RP, Dittus R. Delirium in mechanically ventilated patients: validity and reliability of the confusion assessment method for the intensive care unit (CAM-ICU). JAMA. 2001 Dec 5;286(21):2703-10. doi: 10.1001/jama.286.21.2703. PMID 11730446
- [Background] Mehta S, Cook D, Devlin JW, Skrobik Y, Meade M, Fergusson D, Herridge M, Steinberg M, Granton J, Ferguson N, Tanios M, Dodek P, Fowler R, Burns K, Jacka M, Olafson K, Mallick R, Reynolds S, Keenan S, Burry L; SLEAP Investigators; Canadian Critical Care Trials Group. Prevalence, risk factors, and outcomes of delirium in mechanically ventilated adults. Crit Care Med. 2015 Mar;43(3):557-66. doi: 10.1097/CCM.0000000000000727. PMID 25493968
- [Background] Milbrandt EB, Deppen S, Harrison PL, Shintani AK, Speroff T, Stiles RA, Truman B, Bernard GR, Dittus RS, Ely EW. Costs associated with delirium in mechanically ventilated patients. Crit Care Med. 2004 Apr;32(4):955-62. doi: 10.1097/01.ccm.0000119429.16055.92. PMID 15071384
- [Background] Knauert MP, Gilmore EJ, Murphy TE, Yaggi HK, Van Ness PH, Han L, Hirsch LJ, Pisani MA. Association between death and loss of stage N2 sleep features among critically Ill patients with delirium. J Crit Care. 2018 Dec;48:124-129. doi: 10.1016/j.jcrc.2018.08.028. Epub 2018 Aug 23. PMID 30179762
- [Background] Pandharipande PP, Girard TD, Jackson JC, Morandi A, Thompson JL, Pun BT, Brummel NE, Hughes CG, Vasilevskis EE, Shintani AK, Moons KG, Geevarghese SK, Canonico A, Hopkins RO, Bernard GR, Dittus RS, Ely EW; BRAIN-ICU Study Investigators. Long-term cognitive impairment after critical illness. N Engl J Med. 2013 Oct 3;369(14):1306-16. doi: 10.1056/NEJMoa1301372. PMID 24088092
- [Background] Witlox J, Eurelings LS, de Jonghe JF, Kalisvaart KJ, Eikelenboom P, van Gool WA. Delirium in elderly patients and the risk of postdischarge mortality, institutionalization, and dementia: a meta-analysis. JAMA. 2010 Jul 28;304(4):443-51. doi: 10.1001/jama.2010.1013. PMID 20664045
- [Background] Pandharipande P, Ely EW. Sedative and analgesic medications: risk factors for delirium and sleep disturbances in the critically ill. Crit Care Clin. 2006 Apr;22(2):313-27, vii. doi: 10.1016/j.ccc.2006.02.010. PMID 16678002
- [Background] Trompeo AC, Vidi Y, Locane MD, Braghiroli A, Mascia L, Bosma K, Ranieri VM. Sleep disturbances in the critically ill patients: role of delirium and sedative agents. Minerva Anestesiol. 2011 Jun;77(6):604-12. PMID 21617624
- [Background] Weinhouse GL, Watson PL. Sedation and sleep disturbances in the ICU. Crit Care Clin. 2009 Jul;25(3):539-49, ix. doi: 10.1016/j.ccc.2009.04.003. PMID 19576529
- [Background] Kanji S, Mera A, Hutton B, Burry L, Rosenberg E, MacDonald E, Luks V. Pharmacological interventions to improve sleep in hospitalised adults: a systematic review. BMJ Open. 2016 Jul 29;6(7):e012108. doi: 10.1136/bmjopen-2016-012108. PMID 27473952
- [Background] Weerink MAS, Struys MMRF, Hannivoort LN, Barends CRM, Absalom AR, Colin P. Clinical Pharmacokinetics and Pharmacodynamics of Dexmedetomidine. Clin Pharmacokinet. 2017 Aug;56(8):893-913. doi: 10.1007/s40262-017-0507-7. PMID 28105598
- [Background] Nelson LE, Lu J, Guo T, Saper CB, Franks NP, Maze M. The alpha2-adrenoceptor agonist dexmedetomidine converges on an endogenous sleep-promoting pathway to exert its sedative effects. Anesthesiology. 2003 Feb;98(2):428-36. doi: 10.1097/00000542-200302000-00024. PMID 12552203
- [Background] Alexopoulou C, Kondili E, Diamantaki E, Psarologakis C, Kokkini S, Bolaki M, Georgopoulos D. Effects of dexmedetomidine on sleep quality in critically ill patients: a pilot study. Anesthesiology. 2014 Oct;121(4):801-7. doi: 10.1097/ALN.0000000000000361. PMID 24988068
- [Background] Turan A, Duncan A, Leung S, Karimi N, Fang J, Mao G, Hargrave J, Gillinov M, Trombetta C, Ayad S, Hassan M, Feider A, Howard-Quijano K, Ruetzler K, Sessler DI; DECADE Study Group. Dexmedetomidine for reduction of atrial fibrillation and delirium after cardiac surgery (DECADE): a randomised placebo-controlled trial. Lancet. 2020 Jul 18;396(10245):177-185. doi: 10.1016/S0140-6736(20)30631-0. PMID 32682483
- [Background] Shehabi Y, Howe BD, Bellomo R, Arabi YM, Bailey M, Bass FE, Bin Kadiman S, McArthur CJ, Murray L, Reade MC, Seppelt IM, Takala J, Wise MP, Webb SA; ANZICS Clinical Trials Group and the SPICE III Investigators. Early Sedation with Dexmedetomidine in Critically Ill Patients. N Engl J Med. 2019 Jun 27;380(26):2506-2517. doi: 10.1056/NEJMoa1904710. Epub 2019 May 19. PMID 31112380
- [Background] Su X, Meng ZT, Wu XH, Cui F, Li HL, Wang DX, Zhu X, Zhu SN, Maze M, Ma D. Dexmedetomidine for prevention of delirium in elderly patients after non-cardiac surgery: a randomised, double-blind, placebo-controlled trial. Lancet. 2016 Oct 15;388(10054):1893-1902. doi: 10.1016/S0140-6736(16)30580-3. Epub 2016 Aug 16. PMID 27542303
- [Background] Wu XH, Cui F, Zhang C, Meng ZT, Wang DX, Ma J, Wang GF, Zhu SN, Ma D. Low-dose Dexmedetomidine Improves Sleep Quality Pattern in Elderly Patients after Noncardiac Surgery in the Intensive Care Unit: A Pilot Randomized Controlled Trial. Anesthesiology. 2016 Nov;125(5):979-991. doi: 10.1097/ALN.0000000000001325. PMID 27571256
- [Background] Zhang DF, Su X, Meng ZT, Li HL, Wang DX, Xue-Ying Li, Maze M, Ma D. Impact of Dexmedetomidine on Long-term Outcomes After Noncardiac Surgery in Elderly: 3-Year Follow-up of a Randomized Controlled Trial. Ann Surg. 2019 Aug;270(2):356-363. doi: 10.1097/SLA.0000000000002801. PMID 29742525
- [Background] Skrobik Y, Duprey MS, Hill NS, Devlin JW. Low-Dose Nocturnal Dexmedetomidine Prevents ICU Delirium. A Randomized, Placebo-controlled Trial. Am J Respir Crit Care Med. 2018 May 1;197(9):1147-1156. doi: 10.1164/rccm.201710-1995OC. PMID 29498534
- [Background] Sun YM, Zhu SN, Zhang C, Li SL, Wang DX. Effect of low-dose dexmedetomidine on sleep quality in postoperative patients with mechanical ventilation in the intensive care unit: A pilot randomized trial. Front Med (Lausanne). 2022 Aug 31;9:931084. doi: 10.3389/fmed.2022.931084. eCollection 2022. PMID 36117973
- [Background] Barrett W, Buxhoeveden M, Dhillon S. Ketamine: a versatile tool for anesthesia and analgesia. Curr Opin Anaesthesiol. 2020 Oct;33(5):633-638. doi: 10.1097/ACO.0000000000000916. PMID 32826629
- [Background] Wolff K, Winstock AR. Ketamine : from medicine to misuse. CNS Drugs. 2006;20(3):199-218. doi: 10.2165/00023210-200620030-00003. PMID 16529526
- [Background] Schwenk ES, Viscusi ER, Buvanendran A, Hurley RW, Wasan AD, Narouze S, Bhatia A, Davis FN, Hooten WM, Cohen SP. Consensus Guidelines on the Use of Intravenous Ketamine Infusions for Acute Pain Management From the American Society of Regional Anesthesia and Pain Medicine, the American Academy of Pain Medicine, and the American Society of Anesthesiologists. Reg Anesth Pain Med. 2018 Jul;43(5):456-466. doi: 10.1097/AAP.0000000000000806. PMID 29870457
- [Background] Devlin JW, Skrobik Y, Gelinas C, Needham DM, Slooter AJC, Pandharipande PP, Watson PL, Weinhouse GL, Nunnally ME, Rochwerg B, Balas MC, van den Boogaard M, Bosma KJ, Brummel NE, Chanques G, Denehy L, Drouot X, Fraser GL, Harris JE, Joffe AM, Kho ME, Kress JP, Lanphere JA, McKinley S, Neufeld KJ, Pisani MA, Payen JF, Pun BT, Puntillo KA, Riker RR, Robinson BRH, Shehabi Y, Szumita PM, Winkelman C, Centofanti JE, Price C, Nikayin S, Misak CJ, Flood PD, Kiedrowski K, Alhazzani W. Clinical Practice Guidelines for the Prevention and Management of Pain, Agitation/Sedation, Delirium, Immobility, and Sleep Disruption in Adult Patients in the ICU. Crit Care Med. 2018 Sep;46(9):e825-e873. doi: 10.1097/CCM.0000000000003299. PMID 30113379
- [Background] Feinberg I, Campbell IG. Ketamine administration during waking increases delta EEG intensity in rat sleep. Neuropsychopharmacology. 1993 Aug;9(1):41-8. doi: 10.1038/npp.1993.41. PMID 8397722
- [Background] Duncan WC, Sarasso S, Ferrarelli F, Selter J, Riedner BA, Hejazi NS, Yuan P, Brutsche N, Manji HK, Tononi G, Zarate CA. Concomitant BDNF and sleep slow wave changes indicate ketamine-induced plasticity in major depressive disorder. Int J Neuropsychopharmacol. 2013 Mar;16(2):301-11. doi: 10.1017/S1461145712000545. Epub 2012 Jun 7. PMID 22676966
- [Background] Faraguna U, Vyazovskiy VV, Nelson AB, Tononi G, Cirelli C. A causal role for brain-derived neurotrophic factor in the homeostatic regulation of sleep. J Neurosci. 2008 Apr 9;28(15):4088-95. doi: 10.1523/JNEUROSCI.5510-07.2008. PMID 18400908
- [Background] Song B, Zhu J. A Novel Application of Ketamine for Improving Perioperative Sleep Disturbances. Nat Sci Sleep. 2021 Dec 25;13:2251-2266. doi: 10.2147/NSS.S341161. eCollection 2021. PMID 34992482
- [Background] Duncan WC Jr, Ballard ED, Zarate CA. Ketamine-Induced Glutamatergic Mechanisms of Sleep and Wakefulness: Insights for Developing Novel Treatments for Disturbed Sleep and Mood. Handb Exp Pharmacol. 2019;253:337-358. doi: 10.1007/164_2017_51. PMID 28939975
- [Background] Berman RM, Cappiello A, Anand A, Oren DA, Heninger GR, Charney DS, Krystal JH. Antidepressant effects of ketamine in depressed patients. Biol Psychiatry. 2000 Feb 15;47(4):351-4. doi: 10.1016/s0006-3223(99)00230-9. PMID 10686270
- [Background] Abdallah CG, Adams TG, Kelmendi B, Esterlis I, Sanacora G, Krystal JH. KETAMINE'S MECHANISM OF ACTION: A PATH TO RAPID-ACTING ANTIDEPRESSANTS. Depress Anxiety. 2016 Aug;33(8):689-97. doi: 10.1002/da.22501. Epub 2016 Apr 6. PMID 27062302
- [Background] Newport DJ, Carpenter LL, McDonald WM, Potash JB, Tohen M, Nemeroff CB; APA Council of Research Task Force on Novel Biomarkers and Treatments. Ketamine and Other NMDA Antagonists: Early Clinical Trials and Possible Mechanisms in Depression. Am J Psychiatry. 2015 Oct;172(10):950-66. doi: 10.1176/appi.ajp.2015.15040465. PMID 26423481
- [Background] Kishimoto T, Chawla JM, Hagi K, Zarate CA, Kane JM, Bauer M, Correll CU. Single-dose infusion ketamine and non-ketamine N-methyl-d-aspartate receptor antagonists for unipolar and bipolar depression: a meta-analysis of efficacy, safety and time trajectories. Psychol Med. 2016 May;46(7):1459-72. doi: 10.1017/S0033291716000064. Epub 2016 Feb 12. PMID 26867988
- [Background] Bartova L, Papageorgiou K, Milenkovic I, Dold M, Weidenauer A, Willeit M, Winkler D, Kasper S. Rapid antidepressant effect of S-ketamine in schizophrenia. Eur Neuropsychopharmacol. 2018 Aug;28(8):980-982. doi: 10.1016/j.euroneuro.2018.05.007. Epub 2018 Jul 2. PMID 30041987
- [Background] Molero P, Ramos-Quiroga JA, Martin-Santos R, Calvo-Sanchez E, Gutierrez-Rojas L, Meana JJ. Antidepressant Efficacy and Tolerability of Ketamine and Esketamine: A Critical Review. CNS Drugs. 2018 May;32(5):411-420. doi: 10.1007/s40263-018-0519-3. PMID 29736744
- [Background] Canuso CM, Singh JB, Fedgchin M, Alphs L, Lane R, Lim P, Pinter C, Hough D, Sanacora G, Manji H, Drevets WC. Efficacy and Safety of Intranasal Esketamine for the Rapid Reduction of Symptoms of Depression and Suicidality in Patients at Imminent Risk for Suicide: Results of a Double-Blind, Randomized, Placebo-Controlled Study. Am J Psychiatry. 2018 Jul 1;175(7):620-630. doi: 10.1176/appi.ajp.2018.17060720. Epub 2018 Apr 16. PMID 29656663
- [Background] Segmiller F, Ruther T, Linhardt A, Padberg F, Berger M, Pogarell O, Moller HJ, Kohler C, Schule C. Repeated S-ketamine infusions in therapy resistant depression: a case series. J Clin Pharmacol. 2013 Sep;53(9):996-8. doi: 10.1002/jcph.122. Epub 2013 Jul 24. No abstract available. PMID 23893490
- [Background] Persson J, Hasselstrom J, Maurset A, Oye I, Svensson JO, Almqvist O, Scheinin H, Gustafsson LL, Almqvist O. Pharmacokinetics and non-analgesic effects of S- and R-ketamines in healthy volunteers with normal and reduced metabolic capacity. Eur J Clin Pharmacol. 2002 Feb;57(12):869-75. doi: 10.1007/s002280100353. PMID 11936706
- [Background] Bornemann-Cimenti H, Wejbora M, Michaeli K, Edler A, Sandner-Kiesling A. The effects of minimal-dose versus low-dose S-ketamine on opioid consumption, hyperalgesia, and postoperative delirium: a triple-blinded, randomized, active- and placebo-controlled clinical trial. Minerva Anestesiol. 2016 Oct;82(10):1069-1076. Epub 2016 Jun 21. PMID 27327855
- [Background] Hu ZC, Xu G, Zhang XW, Ma K, Jin JJ, Li PS. [Meta-analysis of the effects of dexmedetomidine combined with ketamine during dressing changes in burn patients]. Zhonghua Shao Shang Za Zhi. 2020 Jun 20;36(6):458-464. doi: 10.3760/cma.j.cn501120-20190327-00145. Chinese. PMID 32594705
- [Background] Lee KH, Lee SJ, Park JH, Kim SH, Lee H, Oh DS, Kim YH, Park YH, Kim H, Lee SE. Analgesia for spinal anesthesia positioning in elderly patients with proximal femoral fractures: Dexmedetomidine-ketamine versus dexmedetomidine-fentanyl. Medicine (Baltimore). 2020 May;99(20):e20001. doi: 10.1097/MD.0000000000020001. PMID 32443302
- [Background] Zhang Y, Cui F, Ma JH, Wang DX. Mini-dose esketamine-dexmedetomidine combination to supplement analgesia for patients after scoliosis correction surgery: a double-blind randomised trial. Br J Anaesth. 2023 Aug;131(2):385-396. doi: 10.1016/j.bja.2023.05.001. Epub 2023 Jun 9. PMID 37302963
- [Background] Tembo AC, Parker V. Factors that impact on sleep in intensive care patients. Intensive Crit Care Nurs. 2009 Dec;25(6):314-22. doi: 10.1016/j.iccn.2009.07.002. Epub 2009 Oct 31. PMID 19880319
- [Background] Blissitt PA. Sleep and Mechanical Ventilation in Critical Care. Crit Care Nurs Clin North Am. 2016 Jun;28(2):195-203. doi: 10.1016/j.cnc.2016.02.002. Epub 2016 Apr 5. PMID 27215357
- [Background] Roche Campo F, Drouot X, Thille AW, Galia F, Cabello B, d'Ortho MP, Brochard L. Poor sleep quality is associated with late noninvasive ventilation failure in patients with acute hypercapnic respiratory failure. Crit Care Med. 2010 Feb;38(2):477-85. doi: 10.1097/CCM.0b013e3181bc8243. PMID 19789439
- [Background] Lewis K, Piticaru J, Chaudhuri D, Basmaji J, Fan E, Moller MH, Devlin JW, Alhazzani W. Safety and Efficacy of Dexmedetomidine in Acutely Ill Adults Requiring Noninvasive Ventilation: A Systematic Review and Meta-analysis of Randomized Trials. Chest. 2021 Jun;159(6):2274-2288. doi: 10.1016/j.chest.2020.12.052. Epub 2021 Jan 9. PMID 33434496
- [Background] Shinall MC Jr, Arya S, Youk A, Varley P, Shah R, Massarweh NN, Shireman PK, Johanning JM, Brown AJ, Christie NA, Crist L, Curtin CM, Drolet BC, Dhupar R, Griffin J, Ibinson JW, Johnson JT, Kinney S, LaGrange C, Langerman A, Loyd GE, Mady LJ, Mott MP, Patri M, Siebler JC, Stimson CJ, Thorell WE, Vincent SA, Hall DE. Association of Preoperative Patient Frailty and Operative Stress With Postoperative Mortality. JAMA Surg. 2020 Jan 1;155(1):e194620. doi: 10.1001/jamasurg.2019.4620. Epub 2020 Jan 15. PMID 31721994
- [Background] Katayama H, Kurokawa Y, Nakamura K, Ito H, Kanemitsu Y, Masuda N, Tsubosa Y, Satoh T, Yokomizo A, Fukuda H, Sasako M. Extended Clavien-Dindo classification of surgical complications: Japan Clinical Oncology Group postoperative complications criteria. Surg Today. 2016 Jun;46(6):668-85. doi: 10.1007/s00595-015-1236-x. Epub 2015 Aug 20. PMID 26289837
- [Background] Austin PC. An Introduction to Propensity Score Methods for Reducing the Effects of Confounding in Observational Studies. Multivariate Behav Res. 2011 May;46(3):399-424. doi: 10.1080/00273171.2011.568786. Epub 2011 Jun 8. PMID 21818162